CLINICAL TRIAL: NCT03626961
Title: The Role of NEWS on Tertiary Intensive Care Discharges
Brief Title: The Role of NEWS on Intensive Care Discharges
Status: Completed | Type: Observational
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Selcuk KAYIR, Medical doctor, Hitit University
Other Study IDs: 1
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Intensive Care
Keywords: NEWS
MeSH Terms: interventions — Patient Readmission; Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- discharge: patients discharged from icu
  Interventions: Other: readmission; Other: discharge
- readmission: patients readmitted icu in 48 hours after icu discharge
  Interventions: Other: readmission; Other: discharge

INTERVENTIONS:
Other: readmission — Readmission after 48 hours
Other: discharge — Discharge

SUMMARY:
To determine the ability of the NEWS at tertiary intensive care unit discharges to predict the development of clinical deterioration.

To determine a cut-off value for NEWS score for early readmission

DETAILED DESCRIPTION:
The Nationaly Early Warning Score (NEWS) is a single score based on the measurement of vital signs and inspired gases by the patient. A higher NEWS indicates severity of illness and risk of adverse outcomes. The use of NEWS values to select the appropriate patients for tertiary ICU discharges has not been tested. Our aim is to test the value of NEWS on discharges tertiary ICU.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Stay higher than 48 hours

Exclusion Criteria:

* Under 18 years old
* Stay lower than 48 hours
* Intoxication
* Exitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical and medical patients who met the criteria of the tertiary stage intensive care unit
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Readmission rate | 48 hours
  Clinical deterioration within 48 hours after ICU transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur Yagan, Assoc.Prof., Study Chair — Hitit universtiy
Locations (1):
- Hitit university, Çorum, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our regulations forbid to share the IPD